CLINICAL TRIAL: NCT02113787
Title: A Clinical Pharmacokinetics Comparing Brand and Generic Topiramate in Epilepsy Patients : A Open-label,Randomised, Three-period Crossover Study
Brief Title: Switchability Study Between Brand and Generic Topiramate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kon Chu, MD,PhD, professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0620140190 (2013-2172)
Record Dates: First submitted 2014-03-19; First posted 2014-04-15 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Epilepsy
Keywords: epilepsy; anticonvulsants; generic drugs
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacokinetic study, topamed (Active Comparator): For pharmacokinetics, blood samples was taken after receiving Topamax 100mg twice a day in first visit day.
  For pharmacokinetics, blood samples was taken after receiving Topamed 100mg twice a day in second visit day.
  For pharmacokinetics, blood samples was taken after receiving Topamax 100mg twice a day in third visit day.
  For pharmacokinetics, blood samples was taken after receiving Topamed 100mg twice a day in third visit day.
  Interventions: Procedure: Pharmacokinetic study
- Pharmacokinetic study, topamax (Active Comparator): For pharmacokinetics, blood samples was taken after receiving Topamed 100mg twice a day in first visit day.
  For pharmacokinetics, blood samples was taken after receiving Topamax 100mg twice a day in second visit day.
  For pharmacokinetics, blood samples was taken after receiving Topamed 100mg twice a day in third visit day.
  For pharmacokinetics, blood samples was taken after receiving Topamax 100mg twice a day in third visit day.
  Interventions: Procedure: Pharmacokinetic study

INTERVENTIONS:
Procedure: Pharmacokinetic study — Patients who are examen pharmacokinetic study after taking Topamax or Topiramate during 7 days

SUMMARY:
The purpose of the study is to prove the bioequivalence of brand and generic topiramate.

DETAILED DESCRIPTION:
Generic antiepileptic drugs (AED) achieve blood concentration similar to the brand AED. However, controversies exist about efficacy and safety of substituting generic AEDs. Because even minor absorption and kinetic differences can elicit a breakthrough seizure in patients who are changed to a generic AED from brand AED. Therefore, more ideal evaluation of interchangeability from the brand AEDs to generic formulation of the same drug is three-way or four-way crossover study, which can evaluate within-subject variability in pharmacokinetic and pharmacodynamic. Investigator designed four-way crossover study aimed to assess bioequivalence of brand and generic topiramate, to measure trough serum level , and to evaluate efficacy, tolerability and side effect of generic topiramate.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* Patients with epilepsy who take by topamax 100mg bid or who need to take topamax 100mg bid

Exclusion Criteria:

* poor compliance
* subjects whose dose of antiepileptic drug are changed during the study
* subjects whose seizure is not well-controlled judged by neurologist
* history of any kind of drug allergy
* pregnancy or nursing
* existing or recent significant disease (cardiac, hepatic, or renal disease, severe diabetes mellitus, sepsis, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
To Measure the Area under the plasma concentration versus time curve, serum trough drug level of generic and brand topiramate through pharmacokinetics study. | [ Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours after taking the brand or generic topiramate during 7 days]
  All comparisons of the drug formulations fulfill the bioequivalence criteria, with all 90% Confidential intervals(CIs) for Cmax, AUC, and Ctrough being within the 80-125% acceptance range.
  Scaling average bioequivalence that the acceptable bioequivalence limits of 90% CI of generic to brand topiramate will be those limits that are within and/or similar to the bioequivalence limits of the 90% CI of Brand to Brand topiramate

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of generic topiramate in subjects with epilepsy | 4weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kon Chu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Bialer M, Midha KK. Generic products of antiepileptic drugs: a perspective on bioequivalence and interchangeability. Epilepsia. 2010 Jun;51(6):941-50. doi: 10.1111/j.1528-1167.2010.02573.x. Epub 2010 Apr 8. PMID 20384761
- [Background] Erickson SC, Le L, Ramsey SD, Solow BK, Zakharyan A, Stockl KM, Harada AS, Curtis B. Clinical and pharmacy utilization outcomes with brand to generic antiepileptic switches in patients with epilepsy. Epilepsia. 2011 Jul;52(7):1365-71. doi: 10.1111/j.1528-1167.2011.03130.x. Epub 2011 Jun 21. PMID 21692778